# **Informed Consent Form**

**TITLE:** A Hybrid Effectiveness-Implementation Study on Weight Gain Prevention Among 2-1-1 Callers

NCT NUMBER: NCT04373434

**IRB APPROVAL DATE:** October 17, 2023

# Emory University Consent to be a Research Subject

Title: A Hybrid Effectiveness-Implementation Study on Weight Gain Prevention among 2-1-1 Callers.

IRB #: 112359

Principal Investigator: Michelle C. Kegler, MPH, DrPH, Professor in Behavioral, Social, and Health Education Sciences;

Director of the Emory Prevention Research Center.

**Funding Source:** Centers for Disease Control and Prevention

### **Introduction and Study Overview**

Thank you for your interest in our research study. We would like to tell you everything you need to think about before you decide to join the study. It is entirely your choice. If you decide to take part, you can change your mind later and withdraw from the study. You do not have to answer any questions that you do not want to answer.

The purpose of this study is to understand your opinions about the Healthy Homes/Healthy Families research study. The study is funded by the CDC.

#### **Procedures**

If you agree to be in the study, we will conduct a one-time interview by telephone or video call. We will ask you about your experience with the Healthy Homes/Healthy Families research study and the healthy actions you chose to work on, as well as your experiences with being able to get healthy foods. The interview will be audio recorded, and will take about 90 minutes.

#### **Risks and Discomforts**

The risks to you are minimal. You may experience some discomfort when talking about the topics that come up as part of the interview. You do not have to answer any questions that you do not wish to answer and you have the right to withdraw at any time. The risk of breach of confidentiality is minimal. The project team will keep all research records confidential by using a study number instead of your name on any study records wherever possible. Your name and other facts that might point to you will not appear in any report or publication from this project.

#### **Benefits**

This study is not designed to benefit you directly. This study is designed to learn more about your experiences in the Healthy Homes/Healthy Families study and the healthy actions you worked on. The results of this study will help improve the Healthy Homes/Healthy Families program.

#### **Compensation**

You will receive a \$40 gift card for participating in this interview.

#### **Confidentiality**

Study records can be opened by court order. They also may be provided in response to a subpoena or a request for the production of documents. Certain offices and people other than the researchers may look at study records. Government agencies and Emory employees overseeing proper study conduct may look at your study records. These offices include the Office for Human Research Protections, the funder, the Emory Institutional Review Board, and the Emory Office of Research Compliance. Emory will keep any research records we create private to the extent we are required to do so by law. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results.

Page 1 of 2 Version Date: 9/6/2023

IRB Form 8/21/2023



## Voluntary Participation and Withdrawal from the Study

You have the right to leave the study at any time without penalty and you may ask that we not use any information that you have already provided. You may refuse to answer any questions that you do not wish to answer.

# **Contact Information**

If you have questions about this study, your part in it, your rights as a research participant, or if you have questions, concerns or complaints about the research you may contact the following:

- Emory Institutional Review Board at 404-712-0720 or 877-503-9797 or irb@emory.edu

# Consent

| Do you have any questions about anything I just said? Were there any parts that seemed unclear? | | | |
|---|---|---|---|
| Do you agree to take part in the study? | | | |
| Participant agrees to participate: Yes | No | | |
| If Yes: | | | |
| Name of Participant | | | |
| Signature of Person Conducting Informed Consent Discussion | | Date | Time |
| Name of Person Conducting Informed Consent Discussion | | | |

Page 2 of 2 Version Date: 9/6/2023